CLINICAL TRIAL: NCT06658756
Title: Implementation of Internet-Based Psychotherapy for Obsessive-Compulsive Disorder (OCD) in Primary Health Care in Two Cities in the State of São Paulo
Brief Title: Implementation of Internet-Based Psychotherapy for OCD in Primary Health Care in Two Cities in the State of São Paulo
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 74835123.7.0000.0068
Record Dates: First submitted 2024-09-04; First posted 2024-10-26 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-08

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Intervention Model Description: It is a pragmatic clinical treatment, randomized-controlled, parallel, open, two-arm trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- I-CBT (Experimental): Internet cognitive-behavioral therapy
  Interventions: Behavioral: internet-CBT
- TU (No Intervention): Treatment as Usual

INTERVENTIONS:
Behavioral: internet-CBT — 10 modules on line of I-CBT for OCD
  Arms: I-CBT

SUMMARY:
The aim of this study is to assess the implementation of Internet-based Cognitive Behavioral Therapy (I-CBT) treatment in a Brazilian sample.

Researchers will compare 140 participants (70 with I-CBT and 70 in usual care to see if the treatment is feasible.

Participants will undergo online treatment for OCD, lasting 10 to 14 weeks.

DETAILED DESCRIPTION:
Obsessive-compulsive disorder (OCD) affects 2 to 3% of the adult population worldwide. The efficacy of pharmacological therapy with IRS and cognitive-behavioral therapy (CBT) is well recognized, but the clinical spectrum of OCD symptoms makes it difficult for patients to engage in sessions outside the home, decreasing treatment adherence. CBT is a psychological intervention increasingly delivered over the internet, with studies showing its efficacy in patients with OCD. The present study aims to verify the efficacy of implementing internet-based psychotherapy (I-CBT) in the context of a developing country, identifying the barriers and facilitators of this implementation. It will be a pragmatic, randomized-controlled, parallel, open-label, two-arm clinical trial. The implementation will be carried out in the cities of Indaiatuba and Jaguariúna, state of São Paulo, in all their Basic Health Units, in which 140 participants will be randomized between the I-CBT and usual treatment (UT) groups. Results will be assessed post-treatment and at 3- and 12-month follow-up. The hypothesis is that I-CBT is an effective and feasible treatment modality for OCD in a large Brazilian sample.

ELIGIBILITY:
Inclusion Criteria:

* primary diagnosis of OCD according to the DSM-5 (American Psychiatric Association, 2013);
* internet access.

Exclusion Criteria:

* acute suicide risk, assessed by a positive response (1, 2 or 3) to item 9 of the PHQ-9 and considered serious (suicidal imminence) in the suicide risk assessment protocol (S-RAP);
* psychotic symptoms;
* dependence on alcohol or other known psychoactive substances;
* recent bereavement;
* significant cognitive impairment;
* terminal illness for clinical reasons (based on their knowledge of the patient);
* illiterate patients or those unable to read (for example, due to severe dyslexia or visual impairment);
* patients without access to the internet or an electronic device to access the treatment platform.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Y-BOCS | From enrollment to the end of treatment at 10 weeks. 3 and 12 months after end of treatment
  Yale Brown Obsessive-Compulsive Scale. (range from 0 to 40). The lower the score on the scale, the lower the severity or the greater the reduction of symptoms.

SECONDARY OUTCOMES:
PHQ-9 | From enrollment to the end of treatment at 10 weeks. 3 and 12 months after end of treatment
  Patient Health Questionnaire-9 (range 0 to 27). The lower the score on the scale, the lower the severity or the greater the reduction of symptoms
GAD-7 | From enrollment to the end of treatment at 10 weeks. 3 and 12 months after end of treatment
  Generalized Anxiety Disorder 7-item (range 0 to 21). The lower the score on the scale, the lower the severity or the greater the reduction of symptoms.

CONTACTS AND LOCATIONS:
Locations (3):
- Brazil (3):
  - Basic Health System, Indaiatuba, São Paulo
  - University of Sao Paulo General Hospital., São Paulo, São Paulo
  - University of Sao Paulo General Hospital, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD will me available starting after publication.
Access Criteria: Upon request from others researchers.

REFERENCES:
- [Background] Andersson E, Enander J, Andren P, Hedman E, Ljotsson B, Hursti T, Bergstrom J, Kaldo V, Lindefors N, Andersson G, Ruck C. Internet-based cognitive behaviour therapy for obsessive-compulsive disorder: a randomized controlled trial. Psychol Med. 2012 Oct;42(10):2193-203. doi: 10.1017/S0033291712000244. Epub 2012 Feb 21. PMID 22348650
- [Background] Andersson G, Cuijpers P, Carlbring P, Riper H, Hedman E. Guided Internet-based vs. face-to-face cognitive behavior therapy for psychiatric and somatic disorders: a systematic review and meta-analysis. World Psychiatry. 2014 Oct;13(3):288-95. doi: 10.1002/wps.20151. PMID 25273302
- [Background] Andersson G, Carlbring P. Internet-Assisted Cognitive Behavioral Therapy. Psychiatr Clin North Am. 2017 Dec;40(4):689-700. doi: 10.1016/j.psc.2017.08.004. Epub 2017 Sep 19. PMID 29080594
- [Background] Cuijpers P, Riper H. & Andersson G. Internet- based treatment of depression. Current Opinion in Psychology 4, 131-135 (2015).
- [Background] Fairburn CG, Patel V. The impact of digital technology on psychological treatments and their dissemination. Behav Res Ther. 2017 Jan;88:19-25. doi: 10.1016/j.brat.2016.08.012. PMID 28110672
- [Background] Fineberg NA, Reghunandanan S, Simpson HB, Phillips KA, Richter MA, Matthews K, Stein DJ, Sareen J, Brown A, Sookman D; Accreditation Task Force of The Canadian Institute for Obsessive Compulsive Disorders. Obsessive-compulsive disorder (OCD): Practical strategies for pharmacological and somatic treatment in adults. Psychiatry Res. 2015 May 30;227(1):114-25. doi: 10.1016/j.psychres.2014.12.003. Epub 2015 Feb 11. PMID 25681005
- [Background] Gentil AF, Lopes AC, Dougherty DD, Ruck C, Mataix-Cols D, Lukacs TL, Canteras MM, Eskandar EN, Larsson KJ, Hoexter MQ, Batistuzzo MC, Greenberg BD, Miguel EC. Hoarding symptoms and prediction of poor response to limbic system surgery for treatment-refractory obsessive-compulsive disorder. J Neurosurg. 2014 Jul;121(1):123-30. doi: 10.3171/2014.2.JNS131423. Epub 2014 Apr 4. PMID 24702323
- [Background] Goodman WK, Price LH, Rasmussen SA, Mazure C, Fleischmann RL, Hill CL, Heninger GR, Charney DS. The Yale-Brown Obsessive Compulsive Scale. I. Development, use, and reliability. Arch Gen Psychiatry. 1989 Nov;46(11):1006-11. doi: 10.1001/archpsyc.1989.01810110048007. PMID 2684084
- [Background] Karyotaki E, Efthimiou O, Miguel C, Bermpohl FMG, Furukawa TA, Cuijpers P; Individual Patient Data Meta-Analyses for Depression (IPDMA-DE) Collaboration; Riper H, Patel V, Mira A, Gemmil AW, Yeung AS, Lange A, Williams AD, Mackinnon A, Geraedts A, van Straten A, Meyer B, Bjorkelund C, Knaevelsrud C, Beevers CG, Botella C, Strunk DR, Mohr DC, Ebert DD, Kessler D, Richards D, Littlewood E, Forsell E, Feng F, Wang F, Andersson G, Hadjistavropoulos H, Christensen H, Ezawa ID, Choi I, Rosso IM, Klein JP, Shumake J, Garcia-Campayo J, Milgrom J, Smith J, Montero-Marin J, Newby JM, Breton-Lopez J, Schneider J, Vernmark K, Bucker L, Sheeber LB, Warmerdam L, Farrer L, Heinrich M, Huibers MJH, Kivi M, Kraepelien M, Forand NR, Pugh N, Lindefors N, Lintvedt O, Zagorscak P, Carlbring P, Phillips R, Johansson R, Kessler RC, Brabyn S, Perini S, Rauch SL, Gilbody S, Moritz S, Berger T, Pop V, Kaldo V, Spek V, Forsell Y. Internet-Based Cognitive Behavioral Therapy for Depression: A Systematic Review and Individual Patient Data Network Meta-analysis. JAMA Psychiatry. 2021 Apr 1;78(4):361-371. doi: 10.1001/jamapsychiatry.2020.4364. PMID 33471111
- [Background] Lenhard F, Andersson E, Mataix-Cols D, Ruck C, Vigerland S, Hogstrom J, Hillborg M, Brander G, Ljungstrom M, Ljotsson B, Serlachius E. Therapist-Guided, Internet-Delivered Cognitive-Behavioral Therapy for Adolescents With Obsessive-Compulsive Disorder: A Randomized Controlled Trial. J Am Acad Child Adolesc Psychiatry. 2017 Jan;56(1):10-19.e2. doi: 10.1016/j.jaac.2016.09.515. Epub 2016 Oct 25. PMID 27993223
- [Background] Marques L, LeBlanc NJ, Weingarden HM, Timpano KR, Jenike M, Wilhelm S. Barriers to treatment and service utilization in an internet sample of individuals with obsessive-compulsive symptoms. Depress Anxiety. 2010 May;27(5):470-5. doi: 10.1002/da.20694. PMID 20455248
- [Background] McKay D, Sookman D, Neziroglu F, Wilhelm S, Stein DJ, Kyrios M, Matthews K, Veale D. Efficacy of cognitive-behavioral therapy for obsessive-compulsive disorder. Psychiatry Res. 2015 Feb 28;225(3):236-46. doi: 10.1016/j.psychres.2014.11.058. Epub 2014 Dec 8. PMID 25613661
- [Background] Menezes P, Quayle J, Garcia Claro H, da Silva S, Brandt LR, Diez-Canseco F, Miranda JJ, Price LN, Mohr DC, Araya R. Use of a Mobile Phone App to Treat Depression Comorbid With Hypertension or Diabetes: A Pilot Study in Brazil and Peru. JMIR Ment Health. 2019 Apr 26;6(4):e11698. doi: 10.2196/11698. PMID 31025949
- [Background] Mewton L, Smith J, Rossouw P, Andrews G. Current perspectives on Internet-delivered cognitive behavioral therapy for adults with anxiety and related disorders. Psychol Res Behav Manag. 2014 Jan 30;7:37-46. doi: 10.2147/PRBM.S40879. eCollection 2014. PMID 24511246
- [Background] Patel SR, Wheaton MG, Andersson E, Ruck C, Schmidt AB, La Lima CN, Galfavy H, Pascucci O, Myers RW, Dixon LB, Simpson HB. Acceptability, Feasibility, and Effectiveness of Internet-Based Cognitive-Behavioral Therapy for Obsessive-Compulsive Disorder in New York. Behav Ther. 2018 Jul;49(4):631-641. doi: 10.1016/j.beth.2017.09.003. Epub 2017 Sep 15. PMID 29937263
- [Background] Richards D, Richardson T. Computer-based psychological treatments for depression: a systematic review and meta-analysis. Clin Psychol Rev. 2012 Jun;32(4):329-42. doi: 10.1016/j.cpr.2012.02.004. Epub 2012 Feb 28. PMID 22466510
- [Background] Ruck C, Lundstrom L, Flygare O, Enander J, Bottai M, Mataix-Cols D, Andersson E. Study protocol for a single-blind, randomised controlled, non-inferiority trial of internet-based versus face-to-face cognitive behaviour therapy for obsessive-compulsive disorder. BMJ Open. 2018 Sep 5;8(9):e022254. doi: 10.1136/bmjopen-2018-022254. PMID 30185575
- [Background] Ruscio AM, Stein DJ, Chiu WT, Kessler RC. The epidemiology of obsessive-compulsive disorder in the National Comorbidity Survey Replication. Mol Psychiatry. 2010 Jan;15(1):53-63. doi: 10.1038/mp.2008.94. Epub 2008 Aug 26. PMID 18725912
- [Background] Skapinakis P, Caldwell DM, Hollingworth W, Bryden P, Fineberg NA, Salkovskis P, Welton NJ, Baxter H, Kessler D, Churchill R, Lewis G. Pharmacological and psychotherapeutic interventions for management of obsessive-compulsive disorder in adults: a systematic review and network meta-analysis. Lancet Psychiatry. 2016 Aug;3(8):730-739. doi: 10.1016/S2215-0366(16)30069-4. Epub 2016 Jun 16. PMID 27318812
- [Background] Stein MB. Public health perspectives on generalized anxiety disorder. J Clin Psychiatry. 2004;65 Suppl 13:3-7. PMID 15384930
- [Background] Torres AR, Lima MC. [Epidemiology of obsessive-compulsive disorder: a review]. Braz J Psychiatry. 2005 Sep;27(3):237-42. doi: 10.1590/s1516-44462005000300015. Epub 2005 Oct 4. Portuguese. PMID 16224614